CLINICAL TRIAL: NCT00854958
Title: The Diagnosis of Oral Allergy Syndrome Through the Use of a Structured Questionnaire
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Isabel Skypala, Director of Rehabilitation and Therapies, Royal Brompton & Harefield NHS Trust
Other Study IDs: 05/Q0404/38
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-02

CONDITIONS: Food Allergy
Keywords: Oral; Allergy; Syndrome; Food; Pollen
MeSH Terms: conditions — Food Hypersensitivity; Hypersensitivity; Syndrome

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
Oral allergy syndrome is a type of food allergy which mainly affects people with springtime hay fever. It is caused by a cross-reaction, between antibodies to pollens, usually birch tree pollen, and allergens in many different plant foods. It is characterised by symptoms of itching and/or swelling in the mouth and/or throat when eating certain fruits vegetables and nuts. Many of the allergens causing OAS are destroyed by heat, making allergy testing using traditional allergen extracts unreliable. Prick testing or challenging with fresh foods is more reliable, but time consuming, inconvenient and largely unavailable. Pilot study results suggest the characteristic symptoms and foods involved in OAS allow accurate diagnosis using clinical history alone, which forms the basis for the hypothesis of this proposal that OAS can be diagnosed accurately by use of a validated questionnaire alone. The diagnostic questionnaire (PFSDQ), revised from the results of the pilot study, will be tested against two reference test methods, the gold standard of oral food challenge, and the 'platinum standard' of diagnosis made by a medical expert based on history, skin prick testing and oral food challenge. This is not an epidemiological study but with no published studies on OAS in a UK population, this study will also provide some information on the prevalence of OAS in those with springtime hayfever in the UK.

ELIGIBILITY:
Inclusion Criteria:

* symptoms of seasonal allergic rhino-conjunctivitis with/without seasonal asthma from March to May

Exclusion Criteria:

* below the age of 18 years, had poorly controlled concomitant asthma (Forced Expiratory Volume in one second (FEV1) <70% predicted), any significant pre-existing medical condition, were pregnant or required β-blocking agents, H1-receptor antagonists or glucocorticosteroids on a continuous basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult subjects aged over 18 years recruited from the general population
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2005-05; Primary Completion 2006-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The validation of the OAS diagnostic questionnaire (PFSDQ) against accepted standard methods of diagnosis. | 18 months

SECONDARY OUTCOMES:
The characterisation of the pollen and aeroallergen sensitivities of those diagnosed with roal allergy syndrome | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Durham, BA, MA, MD,, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton & Harefield NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Skypala IJ, Calderon MA, Leeds AR, Emery P, Till SJ, Durham SR. Development and validation of a structured questionnaire for the diagnosis of oral allergy syndrome in subjects with seasonal allergic rhinitis during the UK birch pollen season. Clin Exp Allergy. 2011 Jul;41(7):1001-11. doi: 10.1111/j.1365-2222.2011.03759.x. Epub 2011 Apr 25. PMID 21518043